CLINICAL TRIAL: NCT00887510
Title: Metabolic Effects of Antihypertensive Drugs
Brief Title: Metabolic Effects of Antihypertensive Drugs on People With Metabolic Syndrome (The MEAD Study)
Acronym: MEAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 650; K23HL086558 (NIH)
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Hypertension
Keywords: Metabolic Syndrome; High Blood Pressure; Abdominal Obesity; Impaired Glucose Tolerance
MeSH Terms: conditions — Hypertension; Metabolic Syndrome; Obesity, Abdominal; Glucose Intolerance | interventions — Hydrochlorothiazide; trandolapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thiazide First (Active Comparator): Participants will receive 25 mg of hydrochlorothiazide (HCTZ) each day for 6 weeks, followed by 25 mg of HCTZ every day plus 4 mg of trandolapril each day for 6 weeks, followed by 4 mg trandolapril each day for 6 weeks.
  Interventions: Drug: Hydrochlorothiazide; Drug: Trandolapril
- Trandolapril First (Active Comparator): Participants will receive 4 mg of trandolapril each day for 6 weeks, followed by 4 mg of trandolapril for 6 weeks plus 25 mg of HCTZ each day for 6 weeks, followed by 25 mg of HCTZ each day for 6 weeks.
  Interventions: Drug: Hydrochlorothiazide; Drug: Trandolapril

INTERVENTIONS:
Drug: Hydrochlorothiazide — 25 mg tablet once daily for 6 weeks
  Other Names:
  HCTZ
Drug: Trandolapril — 4 mg tablet once daily for 6 weeks

SUMMARY:
High blood pressure, also referred to as hypertension, is a blood pressure level of 140/90 mm Hg or higher. Along with lifestyle changes, various medications are currently used to treat people with hypertension. Some of these medications, however, may affect the way the body handles sugar, essentially preventing the body from breaking down sugar and predisposing people to developing diabetes. People who have metabolic syndrome-a condition primarily characterized by an increased waist measurement, abnormal blood lipid levels, hypertension, and high blood sugar levels-are already at risk of developing diabetes. In these people, taking the antihypertensive medications that prevent sugar breakdown may further increase their risk of diabetes. The purpose of this study is to gain an understanding of how people with metabolic syndrome respond to antihypertensive medications that alter the body's ability to break down sugar.

DETAILED DESCRIPTION:
Treatment for hypertension includes lifestyle changes and medications. Examples of some antihypertensive medications include diuretics, beta-blockers, angiotensin-converting enzyme (ACE) inhibitors, angiotensin receptor blockers (ARBs), and vasodilators. Mounting research suggests that certain antihypertensive medications, such as thiazide diuretics, are associated with metabolic disturbances that result in increased glucose intolerance, while other antihypertensive medications, such as ACE inhibitors and ARBs, appear to improve insulin sensitivity and glucose metabolism. The influence of these medications may be especially critical in people with metabolic syndrome, who are already at risk of developing glucose intolerance and diabetes. The purpose of this study is to gain an understanding of how people with metabolic syndrome respond to antihypertensive medications that alter the body's ability to break down sugar. The long-term goal of the study is to determine the best antihypertensive medications for people who have both metabolic syndrome and hypertension so as to prevent or delay the onset of diabetes in this population.

Participation in this study will last 18 weeks and involve four study visits. Participants will be randomly assigned to initially receive 6 weeks of treatment with either hydrochlorothiazide (HCTZ), which is a thiazide diuretic, or trandolapril, which is an ACE inhibitor. Both medications are FDA-approved for treating hypertension. After 6 weeks of treatment, if participants' blood pressure levels are not too low, they will add the second medication so that they are taking both HCTZ and trandolapril for the next 6 weeks, until Week 12. At Week 12, again if participants' blood pressure levels are not too low, they will then take only the second medication for the last 6 weeks. The four study visits will occur at baseline and after each of the three 6-week treatment periods (Weeks 6, 12, and 18). All study visits will include blood pressure and pulse measurements, urine and blood sampling, oral glucose tolerance testing, and questions about diet and exercise habits. The first and last study visits will also include a physical examination and a medical history review. Some of the blood collected during the first study visit will be used for genetic testing. There will be no follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension, defined as systolic blood pressure greater than or equal to 130 but less than 160 mm Hg and diastolic blood pressure greater than or equal to 85 but less than 110 mm Hg
* Must have any two of the following criteria:

  1. Abdominal obesity, defined as a waist circumference greater than 40 inches in men and greater than 35 inches in women
  2. High-density lipoprotein (HDL) cholesterol level of less than 40 mg/dL in men and less than 50 mg/dL in women
  3. Fasting triglycerides greater than or equal to 150 mg/dL
  4. Fasting glucose level of 100-125 mg/dL

Exclusion Criteria:

* Significant hypertension (greater than 160/110 mm Hg)
* Isolated systolic hypertension
* Diseases requiring treatment with diuretics or angiotensin-converting enzyme (ACE) inhibitors
* Cardiovascular disease (history of heart attack, stroke, heart failure)
* Hypersensitivity to HCTZ or ACE inhibitor
* Type 1 or type 2 diabetes
* Hypokalemia
* Peri-menopause (symptom onset within 1 year)
* Pregnant or breastfeeding
* Secondary causes of hypertension
* Current use of antihypertensive medications known to affect glucose homeostasis (e.g., diuretics, beta blockers, corticosteroids, ACE inhibitors, angiotensin receptor blockers [ARBs])

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-05; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda M. Cooper-DeHoff, Pharm D, MS, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from the University of Florida Shands healthcare system between May 2007 and June 2009.
Pre-assignment Details: 24 participants recruited; 24 randomized, 61 excluded (61 did not meet inclusion criteria)
Period: Overall Study
Arm/Group | Thiazide First | Trandolapril First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Thiazide First | Trandolapril First | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (9.6) | 45.7 (10.6) | 44.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Oral Glucose Tolerance Test (OGTT) Area Under Curve (AUC) After Addition of Trandolapril to Hydrochlorothiazide (HCTZ) Compared With Change in OGTT AUC After Addition of HCTZ to Trandolapril
Description: Comparing the change in OGTT AUC rand 1 visit4-visit 3 with rand 2 visit 3-2. This allows for understanding the effects of addition of trandolapril to 12 weeks of HCTZ compared with addition of HCTZ to 12 weeks of trandolapril. This is the primary outcome of the study.
Time Frame: OGTT AUC measured over 120 minutes after receiving study intervention for 18-24 weeks.
Measure: Mean (Standard Deviation); unit: minutes*mg/dl
Arm/Group | Thiazide First | Trandolapril First
Number analyzed (Participants) | 12 | 12
minutes*mg/dl | -472 (2064) | 1571 (2256)

2. Secondary Outcome: Change in Total Adiponectin Level After Addition of Trandolapril to HCTZ Compared With Change in Adiponectin After Addition of HCTZ to Trandolapril
Description: Comparing the change in adiponectin: rand 1 visit4-visit 3 with rand 2 visit 3-2.
  This allows for understanding the effects of addition of trandolapril to 12 weeks of HCTZ compared with addition of HCTZ to 12 weeks of trandolapril.
Time Frame: Over the course of 18 weeks
Measure: Mean (Standard Deviation); unit: mcg/ml
Arm/Group | Thiazide First | Trandolapril First
Number analyzed (Participants) | 12 | 12
mcg/ml | -1.36 (0.96) | 0.42 (1.11)

ADVERSE EVENTS:
Arm/Group | Thiazide First | Trandolapril First
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thiazide First (N=12) | Trandolapril First (N=12)
Sulfuric acid splatter (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Subject suffered a work related sulfuric acid splatter to bilateral lower extremities. The subject underwent elective excision and grafting and was d/c from hospital 3 days later. Unrelated to study. Subject was taking HCTZ at the time of the event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No